CLINICAL TRIAL: NCT06539871
Title: The Role of Ultrasonography in Detecting Additional Peripheral Nerve Injuries Overshadowed by Clinical and Electrodiagnostic Data in Patients With Peripheral Nerve Injury After the February 6, 2023 Earthquake
Brief Title: The Role of Ultrasonography in the Diagnosis of Double Crush Syndrome
Status: Active, not recruiting | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2023.1676
Record Dates: First submitted 2024-07-31; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Double Crush Syndrome; Earthquake; Peripheral Nerve Injuries
Keywords: Double Crush Syndrome; 6, February 2023 Earhquake; Peripheral Nerve Injuries; Electroneuromyography; Ultrasonography
MeSH Terms: conditions — Peripheral Nerve Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Role of Ultrasonography in Detecting Additional Peripheral Nerve Injuries Overshadowed by Clinical and Electrodiagnostic Data in Patients with Peripheral Nerve Injury After the February 6, 2023 Earthquake

DETAILED DESCRIPTION:
In the study, patients with peripheral nerve injuries who were removed from under the rubble during the earthquake were evaluated. Patients were examined clinically and monitored for possible peripheral nerve and plexus damage.

After obtaining the written and verbal consent of the patients, their identity information, height and weight, professions, the city where they were affected by the earthquake, the duration of their stay under the rubble, the surgical treatments applied until the moment of evaluation, and their medical interventions. The treatments they received (such as steroid use), comorbidities and medications they used were recorded. Patients who had not yet had an ENMG examination were evaluated electrophysiologically. ENMG was then performed by a physiatrist who specializes in peripheral nerve ultrasonography.

In addition to ENMG and sonographic examinations, each patient was evaluated with Quick-DASH (disabilities of the arm, shoulder and hand) and lower extremity functional scale (LEFS) questionnaires.

There are eleven questions in the Quick-DASH survey, each organized on a five-point Likert scale. In these questions, situations related to the functions of the hand, shoulder and upper extremity are questioned. The patient is asked to mark 1 point as "no difficulty", 2 points as "mild difficulty", 3 points as "moderate difficulty", 4 points as "extreme difficulty", and 5 points as "not being able to do it at all". The Quick-DASH score is obtained by subtracting one from the ratio of the total score of the marked items to the number of marked items and multiplying the resulting number by twenty-five. A Quick-DASH score between 0 and 20 indicates normal disability, between 21 and 40 indicates mild disability, between 41 and 60 indicates moderate disability, between 61 and 80 indicates severe disability, and >80 indicates very severe disability.

There are twenty questions in the LEFS survey, each organized on a five-point Likert scale. In these questions, the functionality of the lower extremity in daily life is questioned. The patient is asked to mark "extreme strain or inability" as 0 points, "considerable strain" as 1 point, "moderate strain" as 2 points, "some strain" as 3 points, and "no strain" as 4 points. The minimum score that can be obtained from the survey is zero, while the maximum score is eighty. As the score decreases, it means a decrease in functionality.

Basically, Quick-DASH was applied to the patient with upper extremity nerve injury, LEFS was applied to the patient with lower extremity nerve injury, and both questionnaires were applied to the patients with simultaneous nerve injury in the upper and lower extremities.

ENMG

Sensory nerve conduction studies were performed on bilateral upper extremity median, ulnar, lateral and medial antebrachial and radial nerves in all patients referred to our electrophysiology laboratory with a preliminary diagnosis of upper extremity nerve injury. In median nerve sensory nerve conduction studies, recordings were obtained from the first, second and third fingers, and in ulnar nerve sensory nerve conduction studies, recordings were obtained from the fifth finger. Afterwards, motor nerve conduction studies were performed on the median and ulnar nerves. Motor and sensory conduction velocity, amplitude and latency values for the mentioned nerves were recorded.

In needle EMG, resting potentials were evaluated in the deltoid, biceps, triceps, extensor indicis proprius, abductor pollicis brevis, first dorsal interosseous and abductor digiti minimi muscles for the affected side in all patients. After evaluating MUP morphology, duration and amplitudes in voluntary contraction, the interference pattern in full contraction was examined.

In patients referred with a preliminary diagnosis of lower extremity nerve injury, motor nerve conduction studies on bilateral tibial peroneal nerves and sensory nerve conduction studies on the sural nerve were performed. Motor and sensory conduction velocity, amplitude and latency values for the mentioned nerves were recorded.

The muscles to be evaluated in needle EMG will be determined according to the patient's clinic and the course of the examination, and tibialis anterior, peroneus longus and gastrocnemius muscles were routinely examined in all patients. Depending on the course of the examination, the short head of the biceps femoris, vastus lateralis of the quadriceps femoris, and gluteus medius muscles were also included in the examination. First, the resting potentials of these muscles were evaluated, and then the MUP morphology, duration, and amplitudes in voluntary contraction were evaluated, and the interference pattern in full contraction was examined.

USG

In patients, peripheral nerve ultrasonography was used to detect radial, median and ulnar nerves from bilateral upper extremities; In the lower extremities, examination of the sciatic, peroneal and tibial nerves was planned.

The patient was placed in the supine position and the bilateral upper extremities were examined first in the anatomical neutral position. Then, it was planned to obtain positions where each nerve would be best visualized by giving the patient positions as detailed below.

Median Nerve

The median nerve was first imaged in the axial plane just below the retinaculum flexorum from the volar side of the wrist in the resting position. A preliminary evaluation was made in the axial plane along the nerve trace. Areas with signs of nerve damage such as increased diameter, decrease in density, edema around the nerve, and scar were noted and longitudinal images were taken there. The degree of injury was determined in the longitudinal section.

In all patients, whether or not there was evidence of injury in the axial plane, the median nerve was evaluated under the retinaculum flexorum (at the wrist level), between the flexor digitorum superficialis and digitorum, at the pronotorum teres level, at the elbow level, at the midpoint of the elbow and axilla distance, and in the axillary fossa, and the diameter and area in the axial section were evaluated. Measurements were made sonographically. The midpoint between the elbow and axilla was determined using a tape measure. While measurements were taken from the mid-humerus and axilla, an abduction angle of 60 degrees was given to the shoulder. While measurements were taken outside these two levels, the upper extremities were in a neutral position and longitudinal images were obtained at levels with diameter and area differences compared to the opposite extremity and the degree of nerve damage was determined.

Ulnar Nerve

The ulnar nerve was first imaged in an axial section on the volar aspect of the wrist in the resting position, next to the ulnar artery on the pisiform bone. A rapid evaluation was made in the axial section along the nerve trace and the levels with signs of nerve damage were noted. Diameter-area measurements were taken in these regions and the degree of nerve damage was determined using longitudinal images.

Whether or not there was any evidence of injury in the axial section, measurements were made on the bilateral ulnar nerves on the pisiform bone, at the level of separation with the ulnar artery, in the cubital tunnel, at the midpoint of the distance between the elbow and the axilla, and in the axillary fossa. While measurements at the forearm level were made in the neutral position, the upper extremity was positioned in 90 degrees shoulder abduction, 90 degrees elbow flexion and 90 degrees shoulder external rotation for ulnar nerve imaging in the cubital tunnel. Measurements from the middle of the humerus and the axilla were also made in the same position. Longitudinal images were obtained at levels that differed in diameter and area compared to the opposite extremity, and the degree of nerve damage was determined.

Radial Nerve

The radial nerve was first imaged in an axial section on the volar side, mediolateral to the elbow level, in the resting position. After giving off its superficial and deep branches towards the distal, the deep branch was followed in the axial section until it reached the supinator muscle. Then, the nerve was imaged again at the location where the first image was taken, followed proximally in the axial section, and finally imaged in the axilla. During this process, areas with signs of nerve damage were noted and longitudinal images were taken to determine the degree of nerve damage.

With or without evidence of injury in the axial section, the bilateral radial nerve is inside the supinator muscle (PIN), before entering the supinator muscle (PIN), just before giving off its deep and superficial branches at the elbow level, at the midpoint of the distance between the elbow and the spiral groove, at the level of the spiral groove and in the axillary fossa. Diameter and area measurements were made using axial images. The midpoint of the distance between the spiral groove and the elbow was determined using a tape measure.

Images were obtained in a neutral position at the level before the deep and superficial branches of the radial nerve were divided (at the elbow level). The forearm was pronated 90 degrees to visualize PIN without entering the supinator muscle and within the supinator muscle. While measurements between the elbow and axillary fossa were made, the shoulder was 60 degrees of flexion and 60 degrees of abduction; The elbow was flexed to 90 degrees. Longitudinal images were obtained at levels that differed in diameter and area compared to the opposite extremity, and the degree of nerve damage was determined.

Lower extremity peripheral nerve ultrasonographic examination was performed with the patients in the prone position. The sciatic nerve was first visualized just below the gluteal fold, proximal to the femoral region. From this level, the nerve was followed distally and images were taken at the mid-level of the femur. Afterwards, measurements were made for both nerves at the level where the peroneal and tibial nerves separate. After this stage, firstly, images of the peroneal nerve were taken with axial sections at the proximal part of the fibula head, at the level of the fibula head, at the distal part of the fibula head and at the distal part of the cruris. For the tibial nerve, after peroneal nerve separation, axial cross-section images were taken at the proximal popliteal fossa, popliteal fossa, middle of the cruris and medial malleolus levels. The diameter of the nerve was measured and recorded in the images taken at all mentioned levels. During the tracing, when there were findings suggestive of nerve injury in the nerve segment other than these anatomical levels, a separate measurement was made at that level and noted. Longitudinal images were taken in areas where nerve injury was suspected and the degree of nerve damage was determined.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 12-65
* Being buried under rubble in an earthquake
* Patients with suspected peripheral nerve damage and/or plexus damage after history and physical examination
* Volunteering to participate in the study and signing a consent form

Exclusion Criteria:

* Hemodynamic instability
* Presence of a medical condition that is a contraindication to EMG
* Contact isolation
* Open wound

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients included in the study were rescued from under the rubble. Peripheral nerve damage was considered in all patients and they were referred to us. Patients who were not considered to have peripheral nerve damage after physical examination and electrophysiological examinations were not included in the study.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Ultrasonographic measurements | Ultrasonography examination was performed in 4 patients at the end of the 1st month after the earthquake, in 6 patients at the 3rd month, and in 5 patients at the 6th month.
  For patients with nerve damage in the upper extremities, ultrasonographic examination of the median, ulnar and radial nerves from both upper extremities was performed. Median, ulnar and radial nerves were examined from the wrist level to the axilla. Diameter measurements were made from various points and recorded.
  For patients with nerve damage in the lower extremity, ultrasonographic examination of the sciatic, peroneal and tibial nerves was performed. Sciatic, peroneal and tibial nerves were examined from the ankle level to the gluteal fold level. Diameter measurements were made from various points and recorded.
Electroneuromyographic data | ENMG examination was performed in 4 patients at the end of the 1st month after the earthquake, in 6 patients at the 3rd month, and in 5 patients at the 6th month.
  All patients were examined electrophysiologically. Relevant data and electrophysiological diagnoses were recorded.

OTHER OUTCOMES:
Information obtained from the patient | This information was obtained at the time of initial presentation in all patients.
  Demographic data of all patients, the cities where they were affected by the earthquake, the duration of their stay under the rubble, comorbidities, and the treatments (medical or surgical) they received after the earthquake were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ilker Yagci, Principal Investigator — Marmara University
Locations (1):
- Marmara University Pendik Training and Research Hospital, Istanbul, Pendik, Turkey (Türkiye)